CLINICAL TRIAL: NCT04952597
Title: A Phase 2, Multicenter, Randomized, 3-Arm, Open-Label Study to Investigate the Preliminary Efficacy and Safety of the Anti-TIGIT Monoclonal Antibody Ociperlimab (BGB-A1217) Plus Tislelizumab Plus Concurrent Chemoradiotherapy in Patients With Untreated Limited-Stage Small Cell Lung Cancer
Brief Title: Study of Ociperlimab Plus Tislelizumab Plus Chemoradiotherapy in Participants With Untreated Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AdvanTIG-204; CTR20211531 (Other: ChinaDrugTrials); BGB-A317-A1217-204 (Other: BeiGene ID)
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Limited Stage Small Cell Lung Cancer
MeSH Terms: interventions — tislelizumab; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Ociperlimab + Tislelizumab (Experimental): Ociperlimab plus tislelizumab combined with cCRT (at the investigator's discretion) for 4 cycles (each cycle is 28 days), followed by ociperlimab plus tislelizumab
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Concurrent Chemoradiotherapy
- Arm B: Tislelizumab (Experimental): Tislelizumab combined with cCRT (at the investigator's discretion) for 4 cycles, followed by tislelizumab alone
  Interventions: Drug: Tislelizumab; Drug: Concurrent Chemoradiotherapy
- Arm C: Concurrent Chemoradiotherapy (cCRT) (Experimental): cCRT only for 4 cycles at the investigator's discretion
  Interventions: Drug: Concurrent Chemoradiotherapy

INTERVENTIONS:
Drug: Ociperlimab — Ociperlimab 900 milligrams (mg) administered intravenously once every 3 weeks on Day 1 of each cycle
  Other Names: BGB-A1217
  Arms: Arm A: Ociperlimab + Tislelizumab
Drug: Tislelizumab — Tislelizumab 200 mg administered intravenously once every 3 weeks on Day 1 of each cycle
  Other Names: BGB-A317
  Arms: Arm A: Ociperlimab + Tislelizumab; Arm B: Tislelizumab
Drug: Concurrent Chemoradiotherapy — Cisplatin/Carboplatin: Either cisplatin 75 milligrams/meters squared (mg/m2) administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles or carboplatin at a dose of area under the curve (AUC) 5 administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles.
  Etoposide: (100 mg/m2) administered intravenously on Days 1, 2, and 3 of each cycle for 4 cycles
  Thoracic radiation therapy (TRT): once daily fractions for 6 to 7 weeks for a total dose of 60 to 70 units of absorbed dose of ionizing radiation (Gy)

SUMMARY:
This phase 2 trial examined whether the preliminary efficacy and safety of ociperlimab, tislelizumab, and cCRT when used in combination is expected to advance treatment options in the serious unmet medical need population of Limited-Stage Small Cell Lung Cancer (LS-SCLC) participants .

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has pathologically (histologically or cytologically) proven diagnosis of small cell lung cancer
* Has limited-stage disease (stage Tx, T1-T4, N0-3, M0; AJCC staging, 8th edition), and can be safely treated with definitive radiation doses.
* Participant has not received any prior treatment for LS-SCLC.
* Participant has measurable disease as assessed according to RECIST v1.1 that is appropriate for selection as a target lesion for repeat measurement, as determined by local site investigator/radiology review
* ECOG Performance Status ≤ 2 assessed within 7 days before the first administration of study intervention, and must have a life expectancy of ≥ 12 weeks.

Key Exclusion Criteria:

* Mixed small cell lung cancer histology. Note: mixed SCLC with the component of neuroendocrine carcinoma origin is considered eligible
* Have received surgical resection for LS-SCLC
* Any participant for whom the tumor is considered resectable by surgery or stereotactic body radiation therapy/stereotactic ablative radiotherapy should be considered ineligible
* Is expected to require any other form of antineoplastic therapy while on study.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-TIGIT, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways

Note: Other protocol-defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BeiGene, Study Director — Study Director
Locations (33):
- Tennessee Cancer Specialist, Knoxville, Tennessee, United States
- China (27):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Huai An First Peoples Hospital, Huaian, Jiangsu
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Hanzhong Central Hospital, Hanzhong, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy of Sciences (Ningbo No Hospital), Ningbo, Zhejiang
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbukdo
  - Cha Bundang Medical Center, Cha University, Gyeonggido, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu, Gyeongsangbukdo

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Youling Gong, Qingsong Pang, Rong Yu, Zhengfei Zhu, Jiangqiong Huang, Yufeng Cheng, Diansheng Zhong, Hongbo Wu, Seung Soo Yoo, Tracy Dobbs, Zinan Bao, Yunxia Zuo, Boxian Wei, Pu Sun, You Lu; Abstract CT255: AdvanTIG-204: A phase 2, multicenter, randomized, 3-arm, open-label study investigating the preliminary efficacy and safety of ociperlimab (anti-TIGIT) + tislelizumab (anti-PD-1) + concurrent chemoradiotherapy (cCRT) in patients with untreated limited-stage small cell lung cancer (SCLC). Cancer Res 1 April 2024; 84 (7_Supplement): CT255. https://doi.org/10.1158/1538-7445.AM2024-CT255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in multiple study centers in China, South Korea, and the United States.
Groups:
- Arm A: Ociperlimab + Tislelizumab: Ociperlimab plus tislelizumab combined with cCRT (at the investigator's discretion) for 4 cycles (each cycle is 28 days), followed by ociperlimab plus tislelizumab
  Ociperlimab: Ociperlimab 900 milligrams (mg) administered intravenously once every 3 weeks on Day 1 of each cycle
  Tislelizumab: Tislelizumab 200 mg administered intravenously once every 3 weeks on Day 1 of each cycle
  Concurrent Chemoradiotherapy: Cisplatin/Carboplatin: Either cisplatin 75 milligrams/meters squared (mg/m2) administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles or carboplatin at a dose of area under the curve (AUC) 5 administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles.
  Etoposide: (100 mg/m2) administered intravenously on Days 1, 2, and 3 of each cycle for 4 cycles
  Thoracic radiation therapy (TRT): once daily fractions for 6 to 7 weeks for a total dose of 60 to 70 units of absorbed dose of ionizing radiation (Gy)
- Arm B: Tislelizumab: Tislelizumab combined with cCRT (at the investigator's discretion) for 4 cycles, followed by tislelizumab alone
  Tislelizumab: Tislelizumab 200 mg administered intravenously once every 3 weeks on Day 1 of each cycle
  Concurrent Chemoradiotherapy: Cisplatin/Carboplatin: Either cisplatin 75 milligrams/meters squared (mg/m2) administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles or carboplatin at a dose of area under the curve (AUC) 5 administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles.
  Etoposide: (100 mg/m2) administered intravenously on Days 1, 2, and 3 of each cycle for 4 cycles
  Thoracic radiation therapy (TRT): once daily fractions for 6 to 7 weeks for a total dose of 60 to 70 units of absorbed dose of ionizing radiation (Gy)
- Arm C: Concurrent Chemoradiotherapy (cCRT): cCRT only for 4 cycles at the investigator's discretion
  Concurrent Chemoradiotherapy: Cisplatin/Carboplatin: Either cisplatin 75 milligrams/meters squared (mg/m2) administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles or carboplatin at a dose of area under the curve (AUC) 5 administered intravenously once every 3 weeks on Day 1 of each cycle for 4 cycles.
  Etoposide: (100 mg/m2) administered intravenously on Days 1, 2, and 3 of each cycle for 4 cycles
  Thoracic radiation therapy (TRT): once daily fractions for 6 to 7 weeks for a total dose of 60 to 70 units of absorbed dose of ionizing radiation (Gy)
Period: Overall Study
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Started | 41 | 42 | 43
Completed | 28 | 28 | 25
Not Completed | 13 | 14 | 18
Not completed — Death | 12 | 13 | 14
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) Analysis Set includes all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT) | Total
Number analyzed (Participants) | 41 | 42 | 43 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.50) | 59.9 (7.11) | 61.0 (9.54) | 60.5 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 8 | 27
  Male | 31 | 33 | 35 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 41 | 42 | 42 | 125
  White | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Defined as the time from the date of randomization to the date of the first documented disease progression as determined by the investigator per RECIST v1.1 or death from any cause (whichever occurs first)
Time Frame: Up to approximately 2 years
Population: The ITT analysis set includes all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 41 | 42 | 43
Months | 12.6 [8.7 to NA] — NA: Not estimable due to insufficient number of participants with events | 13.2 [8.5 to NA] — NA: Not estimable due to insufficient number of participants with events | 9.5 [8.3 to 14.4]

2. Secondary Outcome: Complete Response Rate (CR)
Description: defined as the percentage of participants who had CR as assessed by the investigator per RECIST v1.1
Time Frame: Up to approximately 2 years
Population: The Intent-To-Treat (ITT) analysis set includes all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 41 | 42 | 43
percentage of participants | 7.3 [1.5 to 19.9] | 9.5 [2.7 to 22.6] | 2.3 [0.1 to 12.3]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: defined as the percentage of participants who had CR or partial response (PR) as assessed by the investigator per RECIST v1.1
Time Frame: Up to approximately 2 years
Population: The Intent-To-Treat (ITT) analysis set includes all randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 41 | 42 | 43
percentage of participants | 85.4 [70.8 to 94.4] | 88.1 [74.4 to 96.0] | 76.7 [61.4 to 88.2]

4. Secondary Outcome: Overall Response Rate (ORR) in the Programmed Death-Ligand 1 (PD-L1) Analysis Set
Description: as for outcome 3
Time Frame: Up to approximately 2 years
Population: The PD-L1 Analysis Set includes all patients who have at least 1 evaluable PD-L1 measurement expressed by Tumor Area Percentage (TAP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 30 | 28 | 32
percentage of participants
  PD-L1 Expression in TAP ( >=1%): number analyzed (Participants) | 14 | 17 | 17
  PD-L1 Expression in TAP ( >=1%) | 85.7 [57.2 to 98.2] | 94.1 [71.3 to 99.9] | 76.5 [50.1 to 93.2]
  PD-L1 Expression in TAP (<1%): number analyzed (Participants) | 16 | 11 | 15
  PD-L1 Expression in TAP (<1%) | 93.8 [69.8 to 99.8] | 81.8 [48.2 to 97.7] | 86.7 [59.5 to 98.3]

5. Secondary Outcome: Overall Response Rate (ORR) in the T Cell Immunoreceptor With Immunoglobulin and ITIM Domain (TIGIT) Analysis Set
Description: as for outcome 3
Time Frame: Up to approximately 2 years
Population: The TIGIT Analysis Set includes all patients who have at least 1 evaluable TIGIT measurement expressed by Immune Cells (IC) percentage.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 33 | 32 | 35
percentage of participants
  TIGIT Expression Level in IC (>=1%): number analyzed (Participants) | 18 | 25 | 16
  TIGIT Expression Level in IC (>=1%) | 88.9 [65.3 to 98.6] | 88.0 [68.8 to 97.5] | 93.8 [69.8 to 99.8]
  TIGIT Expression Level in IC (<1%): number analyzed (Participants) | 15 | 7 | 19
  TIGIT Expression Level in IC (<1%) | 86.7 [59.5 to 98.3] | 100.0 [59.0 to 100.0] | 68.4 [43.4 to 84.4]

6. Secondary Outcome: Duration of Response (DOR)
Description: defined as the time from the date of the first occurrence of a documented objective response to the date of documented disease progression as assessed by the investigator per RECIST v1.1 or death from any cause (whichever occurs first)
Time Frame: Up to approximately 2 years
Population: The ITT analysis set included all randomized participants; only participants with an objective response (CR or PR) were included in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 35 | 37 | 33
Months | 10.1 [6.0 to NA] — Not estimable due to insufficient number of participants with events | 11.5 [6.9 to NA] — Not estimable due to insufficient number of participants with events | 8.2 [5.6 to NA] — Not estimable due to insufficient number of participants with events

7. Secondary Outcome: Overall Survival (OS) in the ITT Analysis Set
Description: Defined as the time from the date of randomization to the date of death due to any cause
Time Frame: Up to approximately 2 years
Population: The Intent-To-Treat (ITT) analysis set includes all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 41 | 42 | 43
months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | NA [19.8 to NA] — Not estimable due to insufficient number of participants with events | NA [20.0 to NA] — Not estimable due to insufficient number of participants with events

8. Secondary Outcome: Overall Survival (OS) in the PD-L1 Analysis Set
Description: defined as the time from the date of randomization to the date of death due to any cause
Time Frame: Up to approximately 2 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 30 | 28 | 32
months
  PD-L1 Expression in TAP (>=1%): number analyzed (Participants) | 14 | 17 | 17
  PD-L1 Expression in TAP (>=1%) | NA [12.2 to NA] — the median OS was not reached in the PD-L1 expression subgroups due to too few events to draw any meaningful conclusions | NA [17.6 to NA] — the median OS was not reached in the PD-L1 expression subgroups due to too few events to draw any meaningful conclusions | NA [16.5 to NA] — the median OS was not reached in the PD-L1 expression subgroups due to too few events to draw any meaningful conclusions
  PD-L1 Expression in TAP (<1%): number analyzed (Participants) | 16 | 11 | 15
  PD-L1 Expression in TAP (<1%) | NA [13.1 to NA] — the median OS was not reached in the PD-L1 expression subgroups due to too few events to draw any meaningful conclusions | NA [7.3 to NA] — the median OS was not reached in the PD-L1 expression subgroups due to too few events to draw any meaningful conclusions | NA [13.3 to NA] — the median OS was not reached in the PD-L1 expression subgroups due to too few events to draw any meaningful conclusions

9. Secondary Outcome: Overall Survival (OS) in the TIGIT Analysis Set
Description: defined as the time from the date of randomization to the date of death due to any cause
Time Frame: Up to approximately 2 years
Population: The TIGIT Analysis Set includes all patients who have at least 1 evaluable TIGIT measurement expressed by immune cells percentage.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 33 | 32 | 35
months
  TIGIT Expression Level in IC (>=1%): number analyzed (Participants) | 18 | 25 | 16
  TIGIT Expression Level in IC (>=1%) | NA [NA to NA] — the median OS was not reached in the TIGIT expression subgroups, due to too few events to draw any meaningful conclusions | NA [NA to NA] — the median OS was not reached in the TIGIT expression subgroups, due to too few events to draw any meaningful conclusions | NA [20.0 to NA] — the median OS was not reached in the TIGIT expression subgroups, due to too few events to draw any meaningful conclusions
  TIGIT Expression Level in IC (<1%): number analyzed (Participants) | 15 | 7 | 19
  TIGIT Expression Level in IC (<1%) | NA [12.0 to NA] — the median OS was not reached in the TIGIT expression subgroups, due to too few events to draw any meaningful conclusions | NA [17.6 to NA] — the median OS was not reached in the TIGIT expression subgroups, due to too few events to draw any meaningful conclusions | NA [13.3 to NA] — the median OS was not reached in the TIGIT expression subgroups, due to too few events to draw any meaningful conclusions

10. Secondary Outcome: Distant Metastasis-free Survival (DMFS)
Description: defined as the time from the date of randomization to the date of the first documented distant metastasis as assessed by the investigator per RECIST v1.1 or death from any cause (whichever occurs first)
Time Frame: Up to approximately 2 years
Population: The Intent-To-Treat (ITT) analysis set includes all randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 41 | 42 | 43
months | 17.9 [9.7 to NA] — Not estimable due to insufficient number of participants with events | 15.3 [9.8 to NA] — Not estimable due to insufficient number of participants with events | 20.0 [8.6 to NA] — Not estimable due to insufficient number of participants with events

11. Secondary Outcome: PFS in the PD-L1 Analysis Set
Description: defined as the time from the date of randomization to the date of the first documented disease progression as determined by the investigator per RECIST v1.1 or death from any cause (whichever occurs first),
Time Frame: Up to approximately 2 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 30 | 28 | 32
months
  PD-L1 Expression in TAP ( >=1%): number analyzed (Participants) | 14 | 17 | 17
  PD-L1 Expression in TAP ( >=1%) | 12.6 [7.8 to NA] — Not estimable due to insufficient number of participants with events | 15.0 [8.5 to NA] — Not estimable due to insufficient number of participants with events | 11.1 [8.1 to NA] — Not estimable due to insufficient number of participants with events
  PD-L1 Expression in TAP (<1%): number analyzed (Participants) | 16 | 11 | 15
  PD-L1 Expression in TAP (<1%) | 10.3 [5.7 to NA] — Not estimable due to insufficient number of participants with events | 14.8 [4.0 to NA] — Not estimable due to insufficient number of participants with events | 14.4 [7.9 to NA] — Not estimable due to insufficient number of participants with events

12. Secondary Outcome: PFS in the TIGIT Analysis Set
Description: as for outcome 11
Time Frame: Up to approximately 2 years
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 33 | 32 | 35
months
  TIGIT Expression Level in IC (>=1%): number analyzed (Participants) | 18 | 25 | 16
  TIGIT Expression Level in IC (>=1%) | 17.9 [9.5 to NA] — Not estimable due to insufficient number of participants with events | 14.3 [7.1 to NA] — Not estimable due to insufficient number of participants with events | 11.2 [8.3 to NA] — Not estimable due to insufficient number of participants with events
  TIGIT Expression Level in IC (<1%): number analyzed (Participants) | 15 | 7 | 19
  TIGIT Expression Level in IC (<1%) | 8.7 [5.5 to 12.6] | NA [8.3 to NA] — Not estimable due to insufficient number of participants with events | 14.4 [7.2 to NA] — Not estimable due to insufficient number of participants with events

13. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v4.03
Time Frame: From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Population: The Safety Analysis Set includes all patients who have received >= 1 dose of any component of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
Number analyzed (Participants) | 41 | 42 | 43
Participants
  Number of Participants with at least one TEAE | 41 | 42 | 43
  Number of participants with at least one SAE | 25 | 20 | 12

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events (AEs): From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment AEs are defined as events that had an onset date or a worsening in severity from baseline (pretreatment) on or after the first dose of study treatment up to 30 days following study treatment discontinuation or initiation of a new anticancer therapy, whichever occurred first.
Arm/Group | Arm A: Ociperlimab + Tislelizumab | Arm B: Tislelizumab | Arm C: Concurrent Chemoradiotherapy (cCRT)
All-Cause Mortality (participants affected / at risk) | 12/41 | 13/42 | 14/43
Serious Adverse Events (participants affected / at risk) | 25/41 | 20/42 | 12/43
Other Adverse Events (participants affected / at risk) | 41/41 | 42/42 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ociperlimab + Tislelizumab (N=41) | Arm B: Tislelizumab (N=42) | Arm C: Concurrent Chemoradiotherapy (cCRT) (N=43)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 3 (3)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (6) | 5 (5) | 3 (4)
Platelet count decreased (Investigations) | 6 (6) | 3 (4) | 4 (5)
White blood cell count decreased (Investigations) | 5 (6) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ociperlimab + Tislelizumab (N=41) | Arm B: Tislelizumab (N=42) | Arm C: Concurrent Chemoradiotherapy (cCRT) (N=43)
Anaemia (Blood and lymphatic system disorders) | 37 (72) | 38 (79) | 38 (48)
Leukopenia (Blood and lymphatic system disorders) | 2 (4) | 3 (11) | 4 (14)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 2 (15) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 4 (10) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (4) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (5) | 11 (11) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 24 (43) | 19 (35) | 13 (20)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 5 (7) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 2 (2) | 7 (7)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastric dilatation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 34 (73) | 32 (81) | 28 (57)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 22 (40) | 29 (67) | 15 (33)
Asthenia (General disorders) | 9 (14) | 3 (3) | 2 (2)
Chest pain (General disorders) | 3 (3) | 6 (6) | 3 (3)
Fatigue (General disorders) | 7 (9) | 13 (16) | 7 (7)
Malaise (General disorders) | 5 (6) | 3 (4) | 5 (6)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 8 (10) | 4 (6) | 5 (5)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (7) | 6 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 17 (17) | 16 (17) | 14 (14)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3)
Tracheal radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (10) | 8 (10) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 9 (12) | 12 (12) | 5 (7)
Blood bilirubin increased (Investigations) | 6 (7) | 2 (3) | 3 (6)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 4 (4) | 1 (1)
Blood creatinine increased (Investigations) | 2 (6) | 6 (7) | 3 (4)
Blood fibrinogen increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 4 (8) | 1 (2)
C-reactive protein increased (Investigations) | 1 (1) | 3 (6) | 0 (0)
Fibrin D dimer increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 4 (5) | 2 (2)
Lymphocyte count decreased (Investigations) | 11 (28) | 5 (9) | 9 (14)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 28 (88) | 31 (67) | 24 (81)
Platelet count decreased (Investigations) | 26 (59) | 24 (47) | 22 (38)
Red blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 8 (11) | 15 (16) | 6 (6)
White blood cell count decreased (Investigations) | 32 (116) | 31 (96) | 26 (87)
Decreased appetite (Metabolism and nutrition disorders) | 21 (37) | 25 (45) | 18 (22)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (3) | 6 (8) | 4 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (11) | 11 (19) | 4 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (13) | 9 (22) | 6 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (5) | 3 (8) | 3 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (22) | 9 (17) | 4 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (6)
Hypochloraemia (Metabolism and nutrition disorders) | 3 (3) | 6 (10) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (12) | 10 (17) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (28) | 21 (37) | 16 (24)
Hypoproteinaemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 6 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (7) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 7 (9) | 3 (4)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 5 (7) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 11 (12) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 3 (3) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (32) | 33 (40) | 33 (35)
Eczema (Skin and subcutaneous tissue disorders) | 5 (7) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 16 (17) | 2 (4) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 5 (7) | 4 (8)
Hypotension (Vascular disorders) | 1 (1) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT04952597/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04952597/SAP_001.pdf